CLINICAL TRIAL: NCT00276354
Title: Tolerance of Long Term Administration of Forlax® 10g in Elderly Ambulatory or Institutionalized Patients Suffering From Chronic Constipation. Single Blind Randomised Lactulose-controlled Study With Individual Expected Benefit.
Brief Title: Study of Long-term Use of Forlax® in Elderly Patients With Chronic Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-31-52072-003
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Polyethylene Glycols

INTERVENTIONS:
Drug: PEG 4000 (Forlax ®)

SUMMARY:
The main purpose of this study is to evaluate the tolerance of long term repeated doses of Forlax® 10g versus lactulose in elderly ambulatory or institutionalized patients, paying special attention to digestive and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized patients (in a medical care ward) for at least 3 months, or ambulatory patients
* Suffering from chronic constipation defined as:

  * either less than 3 stools per week for at least 3 months and no or partial efficacy of dietary advices, OR
  * patient treated with laxative medication/s for at least 3 months before inclusion, because of chronic constipation corresponding to less than 3 stools per week in case of no laxative treatment
* patient has less than 3 stools during 7 consecutive days of the screening wash-out period

Exclusion Criteria:

* known organic intestinal disease
* having had intestinal surgery
* abdominal or pelvic radiation, carcinoma, obstructive disease, malabsorption disease
* fecal mass in the rectum which cannot be completely evacuated during the screening wash-out period

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 246 (Actual)
Dates: Start 1999-12; Study Completion 2001-11-20 (Actual)

PRIMARY OUTCOMES:
Clinical and biological tolerance with special attention to digestive and nutritional status. Clinical tolerance will be assessed by digestive symptomatology collected on a daily basis
Digestive examination assessed at screening wash-out period and each month
Nutritional status assessed at screening wash-out period, month 3 and month 6
Vital signs assessed at screening wash-out period, month 3 and month 6. Biological tolerance will be assessed by nutritional markers, malabsorption markers and routine laboratory tests assessed at screening wash-out period and month 3 and 6.
Drug interaction assessment assessed at screening wash-out period and month 3 and 6.

SECONDARY OUTCOMES:
Long term efficacy based on daily nurse diary
Healthcare cost analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (146):
- France (146):
  - 19 rue Jules Guesde, Abscon
  - Centre Saint Victor, Amiens
  - 117 ter rue Jean Jaurès, Anzin
  - 8 rue Jean Jaurès, Anzin
  - 26 av. Charles de Gaulle, Aubevoye
  - 89 avenue de Niort, Beauvoir-sur-Niort
  - 11 Place de la République, Blois
  - 39, avenue de France, Blois
  - 30 rue Bayeux, Bretteville-l'Orgueilleuse
  - 30 rue Pasteur, Bruille-lez-Marchiennes
  - 6 avenue du 6 Juin, Caen
  - 98 Boulevard du Maréchal Lyautey, Caen
  - Rue de l'Hôtel de Ville, Carquefou
  - La Cerisaie, Castelmaurou
  - 33 rue Gambetta, Château-Renault
  - 94 bis bld de la République, Châtelaillon-Plage
  - 25 avenue de Nantes, Cholet
  - 116 rue Henri Barbusse, Denain
  - 25 Place Gambetta, Denain
  - 6 rue de Ronde, Derval
  - CHS de la Chartreuse, Dijon
  - 10 rue du Soleil Couchant, Dompierre-sur-Mer
  - 19, avenue de la Gare, Droué
  - 5 route de Paris, Écouis
  - 1 rue du Jardin Botanique, Évreux
  - 6 Centre Commercial les Peupliers, Évreux
  - 8 bis rue du Bout du Pont, Faverolles-sur-Cher
  - 9 rue Cure, Fenioux
  - 15 rue Taffin, Fresnes-sur-Escaut
  - 95 rue Jean-Jaurès, Fresnes-sur-Escaut
  - 14 av. Aristide Briand, Gravigny
  - CHU Grenoble, Grenoble
  - Hôpital Charles Foix, Ivry-sur-Seine
  - Résidence, Grand Maison, L'Union
  - 13 rue Balletant, La Ferté-Imbault
  - 62 rue de Lattre, La Forêt-sur-Sèvre
  - 121 rue M. Delage, La Garde
  - 8 Chemin des Vendéens, La Jubaudière
  - 11 place Sainte Anne, La Riche
  - 194 rue Marius Lacroix, La Rochelle
  - 28 rue du Paradis, La Séguinière
  - 215 route de Bretagne, La Verenne
  - 1, rue de l'Egalité, Lamotte-Beuvron
  - 7 rue de Bel Air, Le Cellier
  - 60 rue de la République, Le Neubourg
  - Hôpital Saint Julien, Le Petit-Quevilly
  - Hôpital Saint-Julien, Le Petit-Quevilly
  - 21 Avenue Gabriel Péri, Le Pradet
  - 360 Avenue de la 1ère DFL, Le Pradet
  - 360, avenue de la 1ère DFL, Le Pradet
  - 390 av. de la lère DFL, Le Pradet
  - 46 Place Paul Flamenq, Le Pradet
  - 61 avenue de la lère DFL, Le Pradet
  - 13 rue de la Libération, Les Andelys
  - Maison de Retrate Saint-Jean, Lille
  - 57 rue Dupont de l'Eure, Louviers
  - 9 rue du Chatel, Louviers
  - Bd Clémenceau, Louviers
  - 8 rue Saint Venant, Luynes
  - 1 rue Pavée, Mainneville
  - Centre de Gérontologie, Yvon Lamour, Maniquerville
  - 4 rue de Champagne, Marly
  - 10 rue des Vignes, Ménigoute
  - 94 rue Henri Urbain, Mortagne-du-Nord
  - 25 rue V. Désormeaux, Mûrs-Erigné
  - 181 rue Paul Bellamy, Nantes
  - 101 Boulevard de Doulon, Nantes
  - 63 rue de la Bottière, Nantes
  - 13 av. de la République, Niort
  - 189 Avenue de la Rochelle, Niort
  - 277 av. de la Rochelle, Niort
  - 6 pl. de la Comédie, Niort
  - 24 rue de la Poste, Niort-Souche
  - 30 Boulevard de la Gare, Nort-sur-Erdre
  - 12 place d'Armes, Nueil-sur-Layon
  - 26 Place Pasteur, Onnaing
  - 76 rue des Ormeaux, Oudon
  - 16 rue Aristide Briand, Pacy-sur-Eure
  - Hôpital Pitié Salpétrière, Paris
  - Centre Hospitalier Sud Hôpital Xavier Arnozan, Pessac
  - 14 rue de Valencay, Périgny
  - 14 rue de Valençay, Périgny
  - 3 Rue Nouvelle, Pierrefitte-sur-Sauldre
  - 29 rue Blin, Pont-de-l'Arche
  - 35 bis rue du Général de Gaulle, Pont-de-l'Arche
  - 28 bis route de Niort, Prahecq
  - 7 rue Gambetta, Quarouble
  - 271 rue Henri Durre, Raismes
  - 338 rue Henri Durre, Raismes
  - Hôpital Boisguillaume - CHU de Rouen, Rouen
  - Hôpital Charles Nicolle - Service de Biochimie Médicale, Rouen
  - Hôpital Charles Nicolle - Service de Gastroentérologie et Nutrition, Rouen
  - Centre Hospitalier, Saint-Amand-les-Eaux
  - 30 av. du Gl. de Gaulle, Saint-Avertin
  - Centre de Long Séjour, Saint-Chamond
  - Centre Hospitalier St Chamond, Saint-Chamond
  - 5 rue Saint Nicolas, Saint-Germain-de-Marencennes
  - 1 rue Vanneau, Saint-Jean-de-Liversay
  - Hôpital de Saint Jean de luz, Saint-Jean-de-Luz
  - 34 rue du Poirier, Saint-Macaire-en-Mauges
  - 53 bld du 8 Mai 1945, Saint-Macaire-en-Mauges
  - Les jardins de Rambam, Saint-Orens-de-Gameville
  - Maison de retraite, Saint-Orens-de-Gameville
  - 36 Rue Louise Michel, Saint-Ouen
  - Chemin Vert, Saint-Pierre-des-Échaubrognes
  - Rue du Petit Montrevault, Saint-Pierre-Montlimart
  - Chemin de la Choisière, Saint-Rémy-en-Mauges
  - 27 rue Principale, Saint-Romain-sur-Cher
  - 12, rue Jean Cocteau, Saint-Saulve
  - 1 Allée Jean Restout, Saint-Sébastien-de-Morsent
  - 19 rue de la Mairie, Saint-Vincent-des-Landes
  - 116 bis rue du 14 Juillet, Sainte-Marie-de-Ré
  - 31 bis rue de la République, Sainte-Marie-de-Ré
  - Les Vergers du Château, Solliès-Pont
  - 31 bis rue de la République, Ste Marie En Ré
  - 28 rue Roger Salengro, Thiant
  - 18 rue de la Baronne, Thilouze
  - 1 rue de Bayeux, Tilly-sur-Seulles
  - 121 av. de la Résistance, Toulon
  - 148 Avenue Cuzin, Toulon
  - 355 Avenue Claret, Toulon
  - 535 av. de la Résistance, Toulon
  - 6 bld Noble le Piermone, Toulon
  - 641 rue Sainte Claire Deville, Toulon
  - 641 rue Sainte Deville, Toulon
  - 15 rue Gimelli, Toulon
  - 112 Avenue du Xvème corps, Toulon
  - 2 pl. Martin Bidouré, Toulon
  - 4 pl. Jean Macé, Toulon
  - Capitole Santé, Toulouse
  - Hostellerie Languedocienne, Toulouse
  - Hôpital de la Grave-Casse Lardit, Toulouse
  - Résidence St Simon, Toulouse
  - 3 rue Maryse Bastié, Tours
  - 81 rue Blaise Pascal, Tours
  - 13 rue Ernest Huard, Tours
  - Centre de Gériatrie du Comte Henry, Troyes
  - Centre Hospitalier de Troyes, Troyes
  - 9 rue Beaurepaire, Valanjou
  - 16 rue Anatole France, Valenciennes
  - Résidence Saly - 2 rue S. Lebourg, Valenciennes
  - 200 rue Jean Jaurès, Vieux-Condé
  - 4 rue Beaurepaire, Vihiers
  - Hôpital Paul Brousse, Villejuif
  - 4, Place Jules Verne, Vineuil
  - 85 rue Jean Jaurès, Wallers